CLINICAL TRIAL: NCT06907108
Title: Clinical, Metabolic, Physical, Functional, Biochemical, Quality of Life, and Quality of Sleep Evaluation in Individuals With Metabolic Syndrome After Performing Systemic Vibratory Therapy on an Oscillating/Vibrating Platform
Brief Title: Evaluation of Clinical, Metabolic, and Physical-functional Effects of Systemic Vibratory Therapy in Metabolic Syndrome
Acronym: SVTandMSy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorio de Vibraçoes Mecanicas e Praticas Integrativas (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 54981315.6.0000.5259; RBR-2bghmh (Registry Identifier: Registro Brasileiro de Ensaios Clínicos (REBEC))
Record Dates: First submitted 2025-03-07; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome; Metabolic Syndrome Obesity; Metabolic Syndrome X
Keywords: whole-body vibration; systemic vibratory therapy; systemic vibration therapy; metabolic syndrome; functionality; quality of life; sleep quality; flexibility; blood parameters; anthropometry; body composition; cardiovascular responses; muscle strength; neuromuscular activation; pain level
MeSH Terms: conditions — Metabolic Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed Frequency (FF) (Active Comparator): In the FF group, a frequency of 5Hz, peak-to-peak displacements of 2.5, 5.0, and 7.5 mm, with 1 min of working time with 10s "on" and 50s "off" and 1 min of rest, were used. During the protocol, the individuals performed static and dynamic squats (intercalated days). One minute of vibration and one minute without vibration were performed in each peak-to-peak displacement, which corresponds to one sequence (one series). From the 1st to the 4th session, 3 sequences were performed (totaling 18 minutes); from the 5th to the 8th session, 4 sequences were performed (totaling 24 minutes); and from the 9th to the 12th session, 5 sequences were performed (totaling 30 minutes).
  Interventions: Device: Systemic vibratory therapy
- Varied Frequency (VF) (Active Comparator): In the VF group, frequencies ranged from 5 to16 Hz (increasing 1 Hz with each session), the work time was 1 min and 1 min rest, and the peak-to-peak displacements of 2.5, 5.0, and 7.5 mm. During the protocol, the individuals performed static and dynamic squats (intercalated days). One minute of vibration and one minute without vibration were performed in each peak-to-peak displacement, which corresponds to one sequence (one series). From the 1st to the 4th session, 3 sequences were performed (totaling 18 minutes); from the 5th to the 8th session, 4 sequences were performed (totaling 24 minutes); and from the 9th to the 12th session, 5 sequences were performed (totaling 30 minutes).
  Interventions: Device: Systemic vibratory therapy

INTERVENTIONS:
Device: Systemic vibratory therapy — The interventions were performed on a vibratory platform with side-alternating displacement of the base (Novaplate Fitness Evolution model, DAF Produtos Hospitalares Ltda, São Paulo). The individual was positioned barefoot, with knees flexed at 130º on the base of the vibratory platform. The protocol was performed over a 6-week period with 2 weekly sessions, totaling 12 sessions. The frequency was 5-16Hz according the protocol, and the peak-to-peak displacement was 2.5, 5.0, and 7.5 mm in all sessions. During the protocol, the individuals performed static and dynamic squats, with one static and one dynamic session (interleaved). The variables were evaluated before and after the interventions.

SUMMARY:
Studies have demonstrated a strong relationship between physical inactivity and the presence of cardiovascular risk factors such as hypertension, insulin resistance, diabetes, dyslipidemia, obesity, and metabolic syndrome. On the other hand, regular physical exercise has been recommended to prevent and treat cardiovascular diseases, their risk factors, and other chronic conditions. Systemic vibration therapy (SVT) has been proposed as an alternative exercise modality for this population.

This project aimed to assess clinical, metabolic, physical, functional, biochemical parameters, quality of life, and sleep quality in individuals with metabolic syndrome undergoing whole-body vibration exercises on a vibratory platform.

This study aimed to evaluate clinical, metabolic, physical-functional, biochemical parameters, quality of life, and sleep quality in individuals with MSy undergoing whole-body vibration exercises. Assessments were conducted before and after the intervention and included cardiovascular responses, dyspnea, fatigue, anthropometric measurements (neck, abdominal, hip, arm, and ankle circumferences), body composition, anterior trunk and lumbar spine flexibility, and laboratory analyses (complete blood count, cholesterol profile, triglycerides, creatinine, uric acid, cortisol, glucose, insulin, growth hormone, vitamin D, and other biomarkers). Questionnaires assessed quality of life and sleep. Neuromuscular function, handgrip strength, lower limb isometric dynamometry, joint goniometry, and functional tests were evaluated.

Participants were randomized into two SVT protocol groups: Fixed Frequency (FF) and Variable Frequency (VF). Both protocols were conducted on a vibratory platform with alternating base displacement.

In the FF group, a frequency of 5 Hz was applied, with peak-to-peak displacements of 2.5, 5.0, and 7.5 mm, a work time of 1 minute (10s "on" and 50s "off"), and 1 minute of rest in an upright position. In the VF group, frequencies varied from 5 to 16 Hz (increasing by 1 Hz per session), with a work time of 1 minute and 1 minute of rest, while peak-to-peak displacements remained the same as in the FF protocol. The protocols were performed in static and dynamic squat positions, twice a week, over six weeks, totaling 12 sessions.

It is expected that this vibratory platform intervention can improve clinical, physical, biochemical, and functional parameters, as well as quality of life and sleep quality in individuals with MSy.

DETAILED DESCRIPTION:
For anamnesis, participant data were collected, including age, sex, smoking status, alcohol consumption, presence and type of diabetes mellitus, presence of systemic arterial hypertension, associated comorbidities, medication use, history of COVID-19, and physical inactivity.

Clinical assessments were conducted before and after the 12 sessions of systemic vibratory therapy, including measurements of systemic blood pressure, heart rate, respiratory rate, the BORG scale, the Numeric Pain Scale (NPS), and the Rating of Perceived Exertion (RPE scale - subjective effort perception). Anthropometric measurements were collected, including neck, abdominal, hip, arm, and ankle circumferences, as well as body composition distribution assessed via bioelectrical impedance, anterior trunk flexibility via the sit-and-reach test (FAT), and lumbar spine flexibility via the Schober test.

Laboratory analyses of relevant biomarkers, the HOMA-IR index, and anthropometric indicators were also evaluated. Questionnaires were administered to assess quality of life and sleep quality.

Neuromuscular activity was assessed using surface electromyography, handgrip strength via a manual dynamometer, lower limb isometric dynamometry, joint goniometry, and functional tests. Patients were positioned on the platform base under the supervision of a healthcare professional to perform the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a confirmed diagnosis of Metabolic Syndrome according to the International Diabetes Federation criteria;
* Aged over 45 years,
* Both sexes.

Exclusion Criteria:

* Uncontrolled untreated hypertension, with elevated systemic blood pressure levels (≥180 x 110 mmHg);
* History of a cardiovascular event (myocardial infarction/stroke) in the last 6 months;
* Deep vein thrombosis while taking medication (6 months);
* History of recent surgery on the lower limbs or spine (within 1 year);
* Neurological, rheumatological, or osteomyoarticular disorders;
* Severe or disabling diseases; individuals with metallic prostheses;
* Individuals unable to undergo the proposed assessments and/or interventions;
* Infectious, neurodegenerative, or pulmonary diseases;
* Individuals who discontinued the intervention (more than three consecutive absences from sessions);
* Individuals presenting any contraindication to the vibratory platform.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin (HbA1c) | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Glycated hemoglobin (HbA1c, %) levels were measured in plasma samples collected after an 8-hour fasting period. Unit of Measure: % (for HbA1c).
  Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Lipid Profile and Fasting Blood Glucose | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglyceride levels were measured in serum samples, and fasting blood glucose levels were measured in plasma samples. All measures collected after an 8-hour fasting period.
  Unit of Measure: mg/dL Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Uric Acid Levels | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Serum uric acid levels were measured in serum samples collected after an 8-hour fasting period.
  Unit of Measure: mg/dL. Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Hormonal Biomarkers | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Insulin, and growth hormone (HGH) levels were assessed in serum samples using standard laboratory techniques after an 8-hour fasting period.
  Unit of Measure: ng/mL. Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Metabolic Biomarkers | From enrollment to the end of treatment at 6 weeks.
  Peripheral blood samples were aseptically collected using an intravenous catheter inserted into an antecubital vein. The blood was separated by centrifugation. Serum cortisol levels were assessed in serum samples using standard laboratory techniques after an 8-hour fasting period.
  Unit of Measure: µg/dL. Sample collection was conducted at the Clinical Analysis Laboratory (Cápsula) of PPC-UERJ, always during the same shift, no later than 8:00 AM.
Total Body Water | From enrollment to the end of treatment at 6 weeks.
  The measure of the Total Body Water of the body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment.
  Unit of Measured: in liters (L).
Lean Body Mass, Fat Mass, and Skeletal Muscle Mass | From enrollment to the end of treatment at 6 weeks.
  The measures of body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment. The following body composition components will be measured:
  Lean Body Mass: Measured in kilograms (kg). Fat Mass: Measured in kilograms (kg). Skeletal Muscle Mass: Measured in kilograms (kg).
Body Fat Percentage | From enrollment to the end of treatment at 6 weeks.
  The Body fat percentage of the body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment.
  Unit of measure: Expressed as a percentage (%).
Visceral Fat Area | From enrollment to the end of treatment at 6 weeks.
  The visceral fat area of the body composition will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment.
  Unit of measure: square centimeters (cm²).
Basal Metabolic Rate | From enrollment to the end of treatment at 6 weeks.
  Basal Metabolic Rate will be analyzed using a Tetrapolar Bioelectrical Impedance Analyzer (InBody 370, BIOSPACE, Republic of Korea). The analyzer performs impedance measurements across five body segments (right arm, left arm, trunk, right leg, and left leg) using three different frequencies (5, 50, and 500 kHz), and provides separate body mass readings for each segment. The device provides separate body mass readings for different body segments, being able to estimate the basal metabolic rate. The basal metabolic rate is directly proportional to the weight and amount of muscle. It was calculated from predictive formulas using the results of the body composition, and involves the data of age, sex and physical activity that is entered into the scale.
  Unit of measure: kilocalories per day (kcal/day).
Body Mass Index (BMI) | From enrollment to the end of treatment at 6 weeks.
  Body Mass Index (BMI) is a clinical index that is used in bioimpedance to assess a person's weight. BMI is calculated by dividing the weight (in kg) by the height (in meters) squared.
  Unit of measure: kilograms per square meter (kg/m²).
Waist-to-Hip Ratio (WHR) | From enrollment to the end of treatment at 6 weeks.
  The ratio of the circumference of the waist to the circumference of the hips, used as an indicator of cardiovascular risk. WHR was calculated by dividing the waist circumference in centimeters by the hip circumference. It is an element for the prognosis of cardiovascular events in adults. The cut-off index for cardiovascular risk is less than 0.85 for women and 0.90 for men. The unit of measurement is unitless.
Waist-to-Height Ratio (WHtR) | From enrollment to the end of treatment at 6 weeks.
  The ratio of the circumference of the waist to height, used as an indicator of metabolic and cardiovascular risk. Height was measured using a vertical stadiometer graduated in centimeters and millimeters. Waist circumference was assessed using a tape measure graduated in centimeters and millimeters. The tape measure was placed midway between the iliac crest and the last rib. This anatomical point has the strongest correlation with abdominal adiposity. The values obtained were stratified into three categories: between 0.40 and 0.44 (lowest % fat, below the risk threshold); between 0.45 and 0.50 (moderate risk); between 0.50 and 0.56 (above the risk threshold). The unit of measurement is unitless.
Conicity Index | From enrollment to the end of treatment at 6 weeks.
  Conicity index is a measure of body fat distribution, particularly visceral fat, calculated using body circumference measurements. The C Index (CI) was determined based on the measurement of body mass, height and waist circumference, in meters, representing an indicator of abdominal obesity, and is based on the principle that some people accumulate fat around the abdomen, with the consequent change in body shape. This index is calculated using the formula:
  C Index = waist circumference (m)/(0.109 x (√ body mass (kg)/height (m))). For the classification of cardiovascular risk, values ≥ 1.18 for women and ≥ 1.25 for men are determined. The unit of measurement is unitless.
Anthropometric measures | From enrollment to the end of treatment at 6 weeks.
  Anthropometric measurements, as circumferences were assessed to evaluate the distribution of fat and other physical characteristics. The circumference measurements will be taken at the following sites, measured in centimeters (cm): neck, waist, hip, arm, and ankle.

SECONDARY OUTCOMES:
Functionality | From enrollment to the end of treatment at 6 weeks.
  The Short Physical Performance Battery (SPPB) is a functional performance test that assesses lower limb function and is used for screening the risk of developing future disabilities. It consists of the following tests:
  Static standing balance, Gait speed, and Sit-to-stand. The total SPPB score ranges from zero (worst performance) to 12 points (best performance) and categorically evaluates performance in the tests through three or four scoring classes: three classes: 0-6 points (poor performance), 7-9 points (moderate performance), and 10-12 points (good performance); or four classes: 0-3 points (deficiency/very poor performance), 4-6 points (poor performance), 7-9 points (moderate performance), and 10-12 points (good performance).
Lumbar spine flexibility | From enrollment to the end of treatment at 6 weeks.
  The Schober Test is used to evaluate lumbar spine flexibility. The examiner marks a horizontal line at the level of the posterior-superior iliac spines and a second line 10 cm above the first. The participant then performs forward trunk flexion, and the difference between the measurements in the standing and flexed positions indicates lumbar flexion. This difference is measured in centimeters (cm). A result of 15 cm is considered indicative of good trunk flexibility and lumbar spine mobility.
  Unit of Measure: Centimeters (cm).
Anterior Trunk Flexion Test | From enrollment to the end of treatment at 6 weeks.
  The Anterior trunk flexion test measures the distance between the tip of the middle finger and the floor after the participant performs forward trunk flexion with feet together and knees straight. The result is recorded in centimeters (cm) and uses the distance between the third finger and the floor.
  Unit of Measure: Centimeters (cm).
Health-related quality of life | From enrollment to the end of treatment at 6 weeks.
  Each participant will complete the World Health Organization Quality of Life - Bref Questionnaire (WHOQOL-Bref) before the first and after the last session. The WHOQOL-Bref is a 26-item instrument that produces scores in four domains (physical health, psychological health, social relationships, and environment) and two items related to overall quality of life (QoL) and general health. The response scales, all five-point Likert-type, range from 1 (not at all/never/very dissatisfied/very poor) to 5 (extremely/always/very satisfied/very good). The average score in each domain reflects the individual's perception of their satisfaction in each aspect of their life, relating to their QoL. The higher the score, the better the perception.
Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of treatment at 6 weeks.
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality and disturbances over a one-month period. This questionnaire consists of 19 self-assessment questions and 5 questions to be answered by bed or room partners. The 19 questions are categorized into 7 components, each scored from 0 to 3. These components include subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The scores for each component are summed to produce a global score ranging from 0 to 21, where higher scores indicate poorer sleep quality. A global PSQI score >5 suggests significant difficulties in at least two components or moderate difficulties in more than three components.
  Unit of Measure: Unitless, scale from 0 to 21. Self-reported questionnaires were administered at two-time points (pre- and post-treatment).
Epworth Sleepiness Scale (ESS) | From enrollment to the end of treatment at 6 weeks.
  The Epworth Sleepiness Scale (ESS) consists of 8 self-reported questions and was used to assess self-reported levels of daytime sleepiness. The questionnaire questions are related to daily activities and have a four-point scale (zero indicating "never dozing off" and 3 indicating "strong chance of dozing off"). The questionnaire scores range from zero to 24. Higher total scores are related to greater sleepiness.
  Self-reported questionnaires administered at two time points (pre- and post-treatment).
Mental health | From enrollment to the end of treatment at 6 weeks.
  The Mini Mental State Examination (MMSE) is a screening instrument to assess the domains (spatial and temporal orientation, immediate and recall memory, calculation, language-naming, repetition, comprehension, writing, and copying of drawings). The MMSE is a cognitive screening test that assesses cognitive function and may indicate dementia. The total score ranges from 0 to 30, with scores above 25 indicating normal cognitive function.
  Score Interpretation:
  26-30 points: Normal cognitive function. 21-24 points: Mild cognitive impairment. 10-20 points: Moderate cognitive impairment. Less than or equal to 9 points: Severe cognitive impairment. Low or very low scores: Strong correlation with dementia, but other mental disorders may also affect the result.
Physical activity | From enrollment to the end of treatment at 6 weeks.
  Assessing the level of physical activity is essential to assess an individual's current health conditions and helps to determine which exercises can be part of their routine. This assessment allows the identification of physical and biological limitations, in addition to finding signs of some diseases. Thus, to classify the level of physical activity of the individual, duly validated questionnaires will be used, such as the International Physical Activity Questionnaire (IPAQ), which allows the estimation of the weekly time spent in moderate and vigorous physical activities in different contexts of daily life. The short version will be applied, consisting of 7 open questions, and its information allows the estimation of the time spent per week in different dimensions of physical activity (walking and physical efforts of moderate and vigorous intensity) and physical inactivity (sitting position).
Cardiovascular responses | From enrollment to the end of treatment at 6 weeks.
  Systemic arterial pressure, heart rate, oxygen saturation and respiratory rate. Resting, training, and recovery heart rates: These will be investigated to assess the intensity of physical effort in terms of the percentage of training achieved. Subjective perception of effort: This will be measured using the Modified Borg Scale. Individuals will be asked about their perception of effort during the interventions. The Borg scale is a numerical scale from "0" to "10", where the patient will indicate a score for their level of dyspnea, at the beginning and end of each session, with "0" being no dyspnea and "10" being maximum dyspnea. The risk of cardiovascular diseases will be calculated using this score. The method provides a prediction of the probability of coronary disease in the population evaluated in ten years, according to age group, sex, systolic and diastolic blood pressure values, values of the ratio between total cholesterol and HDL fraction, presence of smoking and diabetes.
Neuromuscular activation | From enrollment to the end of treatment at 6 weeks.
  A surface electromyograph will be used, which consists of a system with eight analog channels (Miotec™, Biomedical Equipments, Porto Alegre, RS, Brazil) that will continuously record biological signals. The surface electrodes will be positioned on the muscles to be evaluated, and a ground electrode will be positioned on a bony prominence. The standardization proposed by the Surface Electromyography for Non-Invasive Muscle Assessment (SENIAM - http://seniam.org/shoulder_location.htm) guideline will be followed. The evaluated electromyographic signals will be processed through the Miotec Suite™ software (Miotec™, Biomedical Equipments, Porto Alegre, RS, Brazil) and the pertinent analyses will be performed.
Muscle strength | From enrollment to the end of treatment at 6 weeks.
  The Lafayette dynamometer (hand grip dynamometers model j00105) will be used. Participants will be seated with their feet on the floor, their arm in adduction and elbow flexed at 90°, their forearm in a neutral position and their wrist extended between 0° and 30°. Three repetitions of maximum grip of 3 seconds will be performed, with a recovery period of 60 seconds between repetitions.
Pain Level | From enrollment to the end of treatment at 6 weeks.
  It is essential to know the participant's pain, and to assess pain, scales such as the visual analogue scale (VAS) will be used, which consists of a ruler divided into eleven equal parts from zero to ten, where the individual is expected to make the equivalence according to the level of their pain through the numerical classification (zero corresponding to the least and ten to the greatest pain).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina Coelho-Oliveira, Principal Investigator — Laboratório de Vibrações Mecânicas e Integrativas - LAVIMPI/UERJ
Locations (1):
- Laboratório de Vibrações Mecânicas e Práticas Integrativas - Policlínica Universitária Piquet Carneiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD supporting the results in publications will be utilized.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Available indefinitely
Access Criteria: Unending

REFERENCES:
- [Background] Coelho-Oliveira AC, Monteiro-Oliveira BB, Goncalves de Oliveira R, Reis-Silva A, Ferreira-Souza LF, Lacerda ACR, Mendonca VA, Sartorio A, Taiar R, Bernardo-Filho M, Sa-Caputo D. Evidence of Use of Whole-Body Vibration in Individuals with Metabolic Syndrome: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2023 Feb 20;20(4):3765. doi: 10.3390/ijerph20043765. PMID 36834459